CLINICAL TRIAL: NCT05522556
Title: Pre-approval Single-patient Expanded Access for Ritlecitinib (PF-06651600)
Status: Available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B798
Record Dates: First submitted 2022-08-26; First posted 2022-08-31 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Alopecia Areata
Keywords: Alopecia Areata (AA); Alopecia; Patchy AA; Alopecia Universalis (AU); Alopecia Totalis (AT); Ophiasis; Eyelash Loss; Eyebrow Loss; Hair Loss
MeSH Terms: conditions — Alopecia Areata; Alopecia; Alopecia universalis

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Ritlecitinib — capsules

SUMMARY:
Provide pre-approval single patient Expanded Access (compassionate use) of Ritlecitinib for patients.

DETAILED DESCRIPTION:
In Expanded Access, treating physicians are the Sponsors. Expanded Access requests from treating physicians may be submitted to www.pfizercares.com. Availability will depend on location and country.

ELIGIBILITY:
Must have ≥ 50% hair loss on scalp due to Alopecia Areata (AA) and be intolerant or have inadequate response to all commonly used AA therapies accessible in the country. Additional eligibility criteria may be required.

Min Age: 12 Years | Sex: All
Age Groups: Child, Adult, Older Adult